CLINICAL TRIAL: NCT04770025
Title: Transcranial Alternating Current Stimulation to Boost the Efficacy of Motivational Interviewing
Brief Title: A Pilot Study of Non-invasive Brain Stimulation to Boost the Efficacy of Psychotherapy in a Community Sample of People Who Drink Alcohol
Acronym: tACS-MI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Mind Research Network (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-010; P30GM122734 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Motivational Interviewing; Transcranial Electrical Stimulation; Alcohol Drinking
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Double-blind proof-of-concept randomized clinical trial
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Providers/Research Assistants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- MI with tACS (Experimental): Motivational interviewing with concurrent active stimulation
  Interventions: Device: High-density transcranial alternating current stimulation; Behavioral: Motivational interviewing
- MI with sham (Sham Comparator): Motivational interviewing with concurrent sham stimulation
  Interventions: Device: Sham stimulation; Behavioral: Motivational interviewing
- MI-only (Active Comparator): Motivational interviewing only, delayed treatment control
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Device: High-density transcranial alternating current stimulation — High-density electrode configuration with transcranial alternating current stimulation in the beta (15-40Hz) frequency range
  Arms: MI with tACS
Device: Sham stimulation — High-density electrode configuration with sham stimulation
  Arms: MI with sham
Behavioral: Motivational interviewing — Motivational interviewing session focused on alcohol use, approximately 30 minutes in length

SUMMARY:
The goal of this small (n=75) proof-of-concept randomized clinical trial is to test the effects of transcranial alternating current stimulation (tACS) during motivational interviewing (MI) sessions with participants who drink at above the low-risk level. Participants will be randomized to receive either MI with active stimulation, MI with sham stimulation, or a delayed treatment group that receives MI with no stimulation. Measures will include brain imaging, alcohol use, cannabis use, risk-taking behavior, emotions, and others. Participants who are randomized to the delayed-treatment group will not receive brain imaging.

DETAILED DESCRIPTION:
This proof-of-concept randomized clinical trial will recruit n=75 people with problematic levels of drinking who are considering treatment for their alcohol use. These participants will be randomized to one of three conditions: a condition that applies active tACS during an MI session (MI+tACS), a condition that applies sham stimulation during an MI session (MI+sham), or a waitlist control condition (MI-only). Only participants the MI+tACS and MI+sham conditions will be included in the brain imaging portion of the study. One month after their intervention session, all participants will report their use of alcohol in the prior 30 days via an online assessment battery. This will allow us to test the effects of tACS on within-session client speech and outcomes.

Participants will have magnetoencephalography (MEG) scans including rest and an alcohol cue task to measure the acute effects of brain stimulation. Participants will also have MRI scans including structure and rest. The Motivational Interviewing Skill Code (MISC 2.5) and the CASAA Application for Coding Treatment Interactions (CACTI) will be used to assess counselor and participant speech in the recorded MI sessions and to ensure that sessions comply with the principles of MI.

ELIGIBILITY:
Inclusion criteria:

* Self-identify as having problem drinking
* Right-handed
* Age 21-60 years
* AUDIT score indicating risky drinking

Exclusion criteria:

* Left-handed or ambidextrous
* Currently engaged in treatment for alcohol use disorder
* Receiving treatment for alcohol use disorder within the prior 12 months
* History of brain injury or neurological diagnosis
* Evidence of current psychosis
* Past-year substance use disorder other than alcohol, marijuana, or nicotine
* Current or history of severe alcohol withdrawal
* MRI/tACS contraindications including pregnancy
* Impaired hearing (psychotherapy using American Sign Language is not possible within the scope of the proposed study)
* Insufficient corrected visual acuity to complete the assessment instruments
* Unable to read/speak English fluently
* Unable to provide valid informed consent

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Heavy drinking days | One month
  Number of heavy drinking days in the prior 30 days

SECONDARY OUTCOMES:
Drinks per drinking day | One month
  Number of drinks per drink day in the prior 30 days
Percent days abstinent | One month
  Percent days abstinent in the prior 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results reported in a peer-reviewed publication, after deidentification (text, tables, figures, and appendices). Session audio recordings will not be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data. A data use agreement will be required, signed by the requesting investigator and their Authorized Organization Representative (AOR)/Signing Official (SO)

DOCUMENTS (2):
  • Informed Consent Form: Informed Consent (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT04770025/ICF_000.pdf
  • Informed Consent Form: Informed Consent - Phase I online-only (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT04770025/ICF_001.pdf